CLINICAL TRIAL: NCT02153255
Title: Dynamic Gait Analysis in Children With Mucopolysaccharidosis Type IVa
Status: Withdrawn | Type: Observational
Why Stopped: Closure of Gait Analysis Laboratory - unable to set up alternative gait laboratory in time for funders
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Saikat Santra, Consultant in Clinical Inherited Metabolic Disorders, Birmingham Women's and Children's NHS Foundation Trust
Other Study IDs: 14/WM/0120
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Mucopolysaccharidosis IV; Morquio A Disease
Keywords: Morquio; Mucopolysaccharidosis; Galactosamine-6-Sulfatase; GALNS
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children With Mucopolysaccharidosis Type IVa

SUMMARY:
Mucopolysaccharidosis Type IVa (MPS IVa, Morquio Disease) is a rare inherited lysosomal storage disorder caused by deficiency of the enzyme galactose-6-sulfatase.

Children with this disease accumulate a chemical called keratan sulphate, which stops their skeletons developing properly. They are very short in stature and many of their joints are unstable. Children with MPS IVa walk in a different way to other people due to a combination of lax ligaments and skeletal problems such as knock-knees.

Human walking involves the coordinated movements of all four limbs. As we walk, the arms swing oppositely to the legs. This movement pattern is very different in children with MPS IVa. This change seems to involve the whole musculoskeletal system and depends on the severity of the disease.

Recent studies in children with MPS IVa describing walking pattern have concentrated solely on the lower or upper limb respectively, and have not looked at the interaction of the upper and lower limbs during walking.

To our knowledge, the mechanics of walking in children with MPS IVa has not been investigated using a dynamic gait analysis tool (using cameras, sensors and electrodes to track the movements of different parts of the body during walking) and we aim to characterise this in a small number of children with MPS IVa and also examine the effects of splinting the wrist upon the walking pattern to see if this simple intervention makes it easier or more difficult for children with MPS IVa to walk.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPS IVa (documented history of reduced leucocyte GALNS enzyme activity relative to the normal range of the laboratory performing the assay AND/OR molecular analysis showing two pathogenic mutations in the GALNS gene)
* Willing and able to provide written assent and parent/legal guardian able to provide written informed consent after the nature of the study has been explained and prior to any research-related procedures
* Between 6 and 18 years of age inclusive
* Willing to perform all study procedures as far as physically possible

Exclusion Criteria:

* Inability to comply with Gait Analysis protocol (e.g. nonambulant)
* Recent orthopaedic surgery that investigator deems might impact on Gait Analysis
* Use of any investigational product or investigational medical device other than BMN110 within 30 days prior to recruitment, or requirement for any investigational agent other than BMN110 prior to completion of all scheduled study assessments
* Concurrent disease or condition that would interfere with study participation or safety
* Any condition that, in the view of the Principal or Subinvestigators, places the subject at high risk of not completing the study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children With Mucopolysaccharidosis Type IVa
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Evidence of abnormal walking pattern and surface EMG activity as assessed by Dynamic Gait Analysis | Within 6 months of recruitment
  Assessment of head, trunk and joint positions during walking using a 12 camera Vicon motion analysis system. Surface EMG analysis using a 16 channel wireless surface electromyographic (sEMG) system. Assessment of lower limb joint moments and powers using Kistler 9281 and AMTI OPT 400600 force plates.

SECONDARY OUTCOMES:
Change in gait pattern over one year | 12 months after first analysis
  Comparison of two gait analysis studies taken 12 months apart
Effect on gait pattern of using wrist splints | Within 6 months of recruitment
  Assessment of repeat gait analysis measurements done at first visit whilst wearing wrist splints
Effect on gait pattern of lower limb surgery | Within 3 and 6 months of any lower limb surgery
  Further gait analysis studies will be done if a child undergoes any lower limb orthopaedic surgery during the study period and compared with pre-surgery analyses

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham Children's Hospital NHS Foundation Trust, Birmingham, West Midlands, United Kingdom